CLINICAL TRIAL: NCT05751720
Title: Effect on Non-Alcoholic Fatty Liver Disease With Advanced Fibrosis in Patients With Type 2 Diabetes Mellitus on Treatment With Gastric Inhibitory Polypeptide / Glucagon Like Peptide-1 Analogue (Tirzpatide)
Brief Title: Effect on Non-Alcoholic Fatty Liver Disease in Patients With Type 2 Diabetes Mellitus With Gastric Inhibitory Polypeptide/Glucagon Like Peptide-1 Analogue
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Adnan Agha (Other)
Responsible Party: Sponsor-Investigator, Dr Adnan Agha, Assistant Professor, Internal Medicine, College of Medicine and Health Sciences, United Arab Emirates University, United Arab Emirates University
Organization: United Arab Emirates University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAEU_CMHS_IM_startup_AA01
Record Dates: First submitted 2023-02-13; First posted 2023-03-02 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; Type 2 Diabetes; Liver Fat
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Fatty Liver

STUDY DESIGN:
Intervention Model Description: Intervention group will receive GLP-1 analogues (subcutaneous Tirzepatide or oral semaglutide).The dose of oral semaglutide will be 3 mg daily for 30 days (initiation) and if dose then increased to 7 mg daily for 6 months while the dose of Tirzepatide is 0.25 mg once weekly for 4 weeks then 0.5 mg once weekly. The blood tests will be done at baseline, 3 months of treatment and at 6 months of treatment. Liver imaging (fibroscan and/or MRI fat measurement) will be done at baseline and at 6 months to see if there is any change.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GLP-1/GIP Arm pre and post intervention (Experimental): The adult patients with type 2 diabetes mellitus attending Tawam Hospital Diabetes clinic, who are identified as having fatty liver disease either via ultrasound or biochemical parameter of NFS.
  We will aim to include minimum 30 patients fulfilling the selection criteria as below. Informed written consent will be obtained . Intervention group will receive GLP-1 analogues (subcutaneous Tirzepatide or oral semaglutide).
  The blood tests will be done at baseline, 3 months of treatment and at 6 months of treatment. Liver imaging (fibroscan and/or MRI fat measurement) will be done at baseline and at 6 months to see if there is any change.The KPa improvement in liver stiffness and total fat estimation pre and post intervention in both groups will assessed
  Interventions: Drug: GIP/GLP-1a

INTERVENTIONS:
Drug: GIP/GLP-1a — The group will receive GLP-1 analogues (subcutaneous Tirzepatide). The dose of Tirzepatide is 0.25 mg once weekly for 4 weeks then 0.5 mg once weekly.

SUMMARY:
Obesity and type 2 Diabetes Mellitus prevalence has doubled in the last 30 years and nearly one fifth of UAE population has Type 2 Diabetes while more than quarter has obesity.

Non-alcoholic fatty liver disease is present in more than 30% of patients with type 2 diabetes and in > 50% patient with obesity

20% of patients with Non-alcoholic fatty liver disease progress to develop non-alcoholic steatohepatitis which can lead to liver failure and hepatocellular carcinoma.

This study aims to use GLP-1 analogue to see effects on liver fat deposition after six months of treatment

There is no current randomised study on treatment of non-alcoholic steatohepatitis in United Arab Emirates population; so once completed this will the first study.

This study will pave the way for developing a treatment pathway for patients with non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Background:

Over the past few decades Non-Alcoholic Fatty liver disease (NAFLD) related non-alcoholic steatohepatitis (NASH) cirrhosis has overtaken all other causes of liver cirrhosis in the developed world, secondary to the rising epidemic of obesity and type 2 Diabetes mellitus. The prevalence of NAFL is estimated at 30% in developed work and nearly one fifth of them NFALD will progress to NASH, 20% of which will develop liver cirrhosis subsequently leading to liver failure and hepatocellular carcinoma (HCC). Annual medical costs directly attributed to NAFLD exceed €35 billion in top European countries (United Kingdom, France, Germany, and Italy) and over $100 billion in the United States, while cost of this in unknown in Middle East. Non-alcoholic fatty liver disease (NAFLD) is defined as fatty infiltration of the liver not related to alcohol excess or other usual causes of hepatic steatosis (e.g. viral or autoimmune hepatitis or secondary to medications) and includes a spectrum ranging from steatosis, steatohepatitis, and fibrosis to cirrhosis; it is now the most common cause of chronic liver disease worldwide. Although most patients with NAFLD may not progress to advanced fibrosis or cirrhosis, due to the high prevalence the number of patients develop cirrhosis is still high and is now a leading indication for liver transplantation in Europe. Global prevalence data for NAFLD suggest that the, Midlle East region has one of the highest prevalence rate of up to 32%.Type 2 diabetes mellitus (T2DM) is an important risk factor for non-alcoholic fatty liver disease (NAFLD) with recent metanalysis showing that the global prevalence of NAFLD among patients with T2DM to be around 55.5% with no specific available data for Emirati population with respects to NAFLD in T2DM patients. Obesity is another well-known risk factor and there is high prevalence of NAFLD in obese patients, with up to 65% of people with grade I-II obesity (BMI = 30-39.9 kg/m2) and in 85% of patients with grade III obesity (BMI = 40-59 kg/m2) having NAFLD.

United Arab Emirates (UAE) has one of the highest prevalence of type 2 Diabetes Mellitus in the world with 16.4% of adult population diagnosed with this condition as per International Diabetes federation. UAE also has the highest prevalence of obesity, doubled from 1989 to 2017, currently ranking among the top 40 countries in the world with estimated prevalence rate of 31.7%, using body mass index (BMI) cut-off of 30 kg/m2. This rate will be substantially higher if newer definition of ethnicity specific BMI cut off for obesity (i.e. > 25 kg/m2 being obese) is used, which is more relevant for Asian population. The presence of both these conditions means UAE is likely to have very high prevalence of NAFLD in patients having both diabetes and obesity.

The gold standard test for identifying NALFD and Non-alcoholic steatohepatitis (NASH) is a liver biopsy. However, liver biopsy is an invasive procedure and is associated with complications. A non-invasive method using Vibration-controlled transient elastography (VCTE) utilizing FibroScan provides a liver stiffness measurement (LSM) expressed in kilopascals (kPa) which correlate with fibrosis advanced stages like F3 (bridging fibrosis) with LSM of 9.9-13.9 KPa and F4 (advanced scarring or cirrhosis) quite well and has emerged as an alternative to invasive liver biopsy. Other non-invasive tools used to detect the presence of advanced fibrosis in NAFLD include clinical/biochemical scoring systems like NAFLD fibrosis score (NFS) and FIB-4 index, aspartate aminotransferase (AST) to platelet ratio index (APRI), Enhanced Liver Fibrosis panel, Hepascore; and imaging techniques like VCTE or magnetic resonance elastography(MRE). The NFS is based on six clinical/biochemical variables including age, presence of impaired fasting glucose or Diabetes, Body Mass Index (BMI), platelet count, albumin and AST/ALT (alanine aminotransferase) ratio. A recent large meta-analysis, showed that NFS had an area under the receiver operating curve (AUROC) of 0.85 for predicting advanced fibrosis stages like F3 (bridging fibrosis) and F4 (advanced scarring or cirrhosis) with a score of 0.676 or more having 67% sensitivity and 97% specificity to identify the presence of advanced fibrosis. A recent study that compared various risk scores and elastography (including MRE and VCTE) versus liver histology to identify NAFLD fibrosis showed that NFS were better than other indices such as BARD, APRI, and AST/ALT ratio; and found to be as good as MRE and and FIB-4 for predicting advanced fibrosis in patients with biopsy-proven NAFLD. Recent guidelines therefore recommend NFS as a clinically useful tool for identifying patients with NAFLD with a higher likelihood of having advanced fibrosis (F3 or F4).

Currently various treatments have been used for NALFD. The current guidelines from American Association for study of liver diseases suggests that Pioglitazone can improve histological appearance in patient with type 2 Diabetes Mellitus and NASH while Vitamin E may offer benefit in non-diabetic population, while GLP-1 Analgoues like liraglutide could be beneficial however there is not enough evidence for it to be used routinely for patients with NASH.

There is no current data on use of Tirzepatide with NAFLD in Emirati population. There is no literature, to the best of authors knowledge. This study offers our centre and UAE university to be first in the world to trial this study without any known risks and publish new and unique data.

The aim of this study to assess the effects of GLP-1 analogues (subcutaneous Tirzepatide or oral semaglutide) in reducing the fat content and Liver stiffness (using non-invasive imaging methods) in patients with established advanced liver fibrosis with type 2 Diabetes Mellitus in local population.

Specific Aims:

Primary Aim:

To see if GLP-1 analogue causes reduction in liver fat on imaging in patient with type 2 Diabetes Mellitus and NAFLD in our population

Secondary Aims To assess any changes in liver function tests/biochemical profile To see improvement in in NAFLD fibrosis score and it relation to liver fat measurement To see improvement in physical parameters such as weight, BMI, blood pressure To see improvement in blood glucose, HbA1c To assess any reported side effects or tolerability of this combination in local population

Methods, Specific Tasks and Time Schedule:

STUDY DESIGN It is Prospective open label randomized study of adult patients with type 2 diabetes mellitus attending Tawam Hospital Diabetes clinic meeting the selection criteria as below

DATA COLLECTION:

The adult patients with type 2 diabetes mellitus attending Tawam Hospital Diabetes clinic, who are identified as having fatty liver disease either via ultrasound or biochemical parameter of NFS. . The NAFLD fibrosis score (NFS) will be calculated using the published formula (available at website http://gihep.com/calculators/hepatology/nafld-fibrosis-score/).

The investigators will aim to include minimum 30 patients fulfilling the selection criteria as below. Informed written consent will be obtained and the group will receive GLP-1 analogues (subcutaneous Tirzepatide or oral semaglutide). The dose of oral semaglutide will be 3 mg daily for 30 days (initiation) and if dose then increased to 7 mg daily for 6 months while the dose of Tirzepatide is 0.25 mg once weekly for 4 weeks then 0.5 mg once weekly. The blood tests will be done at baseline, 3 months of treatment and at 6 months of treatment. Liver imaging (fibroscan and/or MRI fat measurement) will be done at baseline and at 6 months to see if there is any change.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18; either male or female
* Diagnosed to have Type 2 Diabetes Mellitus for > 1 year.
* Presence of NAFLD advanced fibrosis (F3 and F4; defined by NFS of > 0.676)
* Able to consent independently
* Not already on GLP-1 analogues or SGLT2 inhibitors or pioglitazone
* Good general health
* BMI> 19 but less than 40

Exclusion Criteria:

* Known history of alcohol excess or current alcohol use of > 20 g/week
* Evidence of pre-existing liver or biliary disease (hepatoma, biliary tract obstruction; liver cirrhosis secondary to viral infection or immune/ congenital).
* Known or suspected hypersensitivity to GLP-1 analogues or pioglitazone.
* Receipt of any investigational medicinal product within 30 days before screening.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive methods.
* Endocrinopathies (e.g., Cushing syndrome)
* Personal history of heart disease especially heart failure
* History of malignant neoplasm within 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ is allowed.
* eGFR < 30
* history of heamturia or bladder cancer
* history of osteoporosis
* ALT ≥3.5 times the upper normal limit (UNL)
* Taking steroids, antipsychotics or progesterone preparations
* Uncontrolled hypertension
* Positive insulinoma associated-protein 2 (IA-2) antibodies or anti-glutamic acid decarboxylase (anti-GAD) antibodies.
* HbA1c > 10%
* Claustrophobia or unable to get MRI due to contraindications (e.g metal in the body)
* Weight > 150 kg (due to imaging trolley restrictions)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
change in liver stiffness in terms of kPa | 12 months
  To measure the liver stiffness pre and post GLP-1 analogue/GIP treatment for 6 months to assess any change in liver stiffness in terms of kPa in patient with type 2 Diabetes Mellitus and NAFLD
Change in Liver fat quantification | 12 months
  To measure the liver fat quantification via MRI proton density fraction, pre and post GLP-1 analogue/GIP treatment for 6 months to assess any change in total liver fat content in patients with type 2 Diabetes Mellitus and NAFLD

SECONDARY OUTCOMES:
change in BMI | 12 months
  To measure the body mass index (weight in Kg and height in metres will be combined to report BMI in kg/m2), pre and post GLP-1 analogue/GIP treatment for 6 months to assess any change in BMI in patients with type 2 Diabetes Mellitus and NAFLD
Glycaemic control | 12 months
  To measure the HbA1c, pre and post GLP-1 analogue/GIP treatment for 6 months to assess any change in HbA1c in patients with type 2 Diabetes Mellitus and NAFLD

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Agha, FRCP, Principal Investigator — United Arab Emirates University, College of Medicine & Health Sciences
Locations (1):
- Internal Medicine, College of Medicine and Health Sciences, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Imajo K, Kessoku T, Honda Y, Tomeno W, Ogawa Y, Mawatari H, Fujita K, Yoneda M, Taguri M, Hyogo H, Sumida Y, Ono M, Eguchi Y, Inoue T, Yamanaka T, Wada K, Saito S, Nakajima A. Magnetic Resonance Imaging More Accurately Classifies Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease Than Transient Elastography. Gastroenterology. 2016 Mar;150(3):626-637.e7. doi: 10.1053/j.gastro.2015.11.048. Epub 2015 Dec 8. PMID 26677985
- [Background] Kaswala DH, Lai M, Afdhal NH. Fibrosis Assessment in Nonalcoholic Fatty Liver Disease (NAFLD) in 2016. Dig Dis Sci. 2016 May;61(5):1356-64. doi: 10.1007/s10620-016-4079-4. Epub 2016 Mar 26. PMID 27017224